CLINICAL TRIAL: NCT01457950
Title: A Six Month Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study With a Six Month Open-Label Extension to Evaluate the Efficacy and Safety of Denosumab in Korean Postmenopausal Women With Osteoporosis
Brief Title: A Study in Korean Postmenopausal Women With Osteoporosis to Evaluate the Efficacy and Safety of Denosumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114163
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-02

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: denosumab; Republic of Korea; dual energy x-ray absorptiometry
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): denosumab 60mg subcutaneous injection, single dose at the start of the 6-month double-blind phase
  Interventions: Drug: denosumab
- Arm 2 (Placebo Comparator): placebo subcutaneous injection, single dose at the start of the 6-month double-blind phase
  Interventions: Drug: placebo
- Arm 3 (Experimental): open-label phase follows the double-blind phase, denosumab 60mg subcutaneous injection, single dose at the start of the 6-month open-label phase
  Interventions: Drug: open-label denosumab

INTERVENTIONS:
Drug: denosumab — double-blind phase: 60mg subcutaneous injection, single dose
  Arms: Arm 1
Drug: placebo — double-blind phase: placebo subcutaneous injection, single dose
  Arms: Arm 2
Drug: open-label denosumab — open-label phase: 60mg subcutaneous injection, single dose
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine if denosumab is effective in increasing bone mineral density at the lumbar spine in Korean postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory Korean postmenopausal women with osteoporosis
* greater than 5 years postmenopausal
* aged 60 to 90 years old
* absolute bone mineral density value consistent with a T-score less than -2.5 and greater than or equal to - 4.0 at the either the lumbar spine or total hip, as measured by dual energy x-ray absorptiometry. Subjects with a T-score less than -4.0 are at very high risk for fracture and will be excluded.

Exclusion Criteria:

* previous or current metabolic bone disease, Paget's or Cushing's disease, or hyperprolactinemia
* current hypo- or hyperparathyroidism or hypo- or hyperthyroidism unless on stable thyroid replacement therapy and TSH level meets criteria
* rheumatoid arthritis
* cirrhosis of the liver or unstable liver disease or ALT or AST greater than or equal to 2.0 times the upper limit of normal, or alkaline phosphatase and bilirubin greater than or equal to 1.5 times the upper limit of normal
* medications used to treat osteoporosis, defined for type and duration of use, and including IV and oral bisphosphonates
* medications that affect bone metabolism including parathyroid hormone or derivatives; anabolic steroids or testosterone; glucocorticosteroids; systemic hormone replacement therapy; selective estrogen receptor modulators; tibolone, calcitonin, and calcitriol or vitamin D derivatives; other bone active drugs including anticonvulsives (but not benzodiazepines) and heparin; chronic systemic ketoconazole, androgens, ACTH, cinacalcet, aluminum, lithium, protease inhibitors, methotrexate, and gonadotropin-releasing hormone agonists
* malignancy within 5 years except certain resected types
* malabsorption syndrome or gastrointestinal disorders associated with malabsorption
* abnormal calcium level
* vitamin D deficiency
* any laboratory abnormality that will prevent the subject from completing the study or interfere with interpretation of study results
* severe renal impairment or on dialysis
* impaired immune system or subject is taking immunosuppressants
* oral or dental conditions including current or past history of osteomyelitis or osteonecrosis of the jaw; active dental or jaw condition with requires oral surgery; planned invasive dental procedure; un-healed dental or oral surgery
* any disorder that compromises the ability of the subject to give written informed consent or to comply with study procedures
* any physical or psychiatric disorder that will prevent the subject from completing the study or interferes with study results
* known to have tested positive for HIV
* less than two lumbar vertebrae evaluable for DXA measurements
* height, weight, or girth that may preclude accurate DXA measurements
* drug or alcohol abuse within 12 months that interferes with understanding or completing the study
* known sensitivity to mammalian cell-derived drug products
* use of an investigational drug or device within 30 days of enrollment or currently receiving other investigational agent(s)

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul
  - GSK Investigational Site, Suwon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of a screening phase of up to 2.5 months, a six-month Double-Blind Treatment Phase and a six-month Open-Label Extension Phase. 371 participants (par.) were screened, 135 par. entered the Double-Blind Treatment Phase, and 123 par. continued into the Open-Label Extension Phase.
Groups:
- Denosumab 60 mg: Participants received a denosumab 60 milligrams (mg) single subcutaneous (SC) injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 International Units [IU]).
- Placebo: Participants received a matching placebo single SC injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU).
- Denosumab 60 mg to Open-Label Denosumab 60mg: Participants received a denosumab 60 milligrams (mg) single subcutaneous (SC) injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 International Units [IU]). At the end of the Double-Blind Treatment Phase, following completion of all Month 6 assessments, eligible participants entered the Open-Label Extension Phase and received a single SC injection of denosumab 60 mg and were followed up for an additional 6 months.
- Placebo to Open-Label Denosumab 60 mg: Participants received a matching placebo single SC injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU). At the end of the Double-Blind Treatment Phase, following completion of all Month 6 assessments, eligible participants entered the Open-Label Extension Phase and received a single SC injection of denosumab 60 mg and were followed up for an additional 6 months.
Period: Double-Blind Phase
Arm/Group | Denosumab 60 mg | Placebo | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Started | 69 | 66 | 0 | 0
Completed the 6 Month Assessment | 62 ("Completed 6 month assessment" refers to par. that completed at least one 6 month assessment.) | 64 ("Completed 6 month assessment" refers to par. that completed at least one 6 month assessment.) | 0 | 0
Completed | 60 ("Completed" refers to par. that did not have a withdraw reason at the 6 month visit.) | 63 ("Completed" refers to par. that did not have a withdraw reason at the 6 month visit.) | 0 | 0
Not Completed | 9 | 3 | 0 | 0
Not completed — Continuation Criteria Not Met | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 0 | 0
Period: Open-Label Phase
Arm/Group | Denosumab 60 mg | Placebo | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Started | 0 | 0 | 60 | 63
Completed | 0 | 0 | 58 | 61
Not Completed | 0 | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg | Placebo | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (4.86) | 66.0 (4.77) | 66.5 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 66 | 135
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Lumbar Spine BMD at Month 6
Description: Mean percent change from Baseline in lumbar spine bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using the Analysis of Covariance (ANCOVA) model adjusting for treatment and Baseline BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Baseline=(measure at Month 6 - measure at Baseline) divided by the measure at Baseline * 100.
Time Frame: Baseline and Month 6
Population: Intent-to-Treat Efficacy (ITTE) Population: all participants who received one dose of study medication, and had a Baseline measure and at least one post-Baseline efficacy measure during the Double-Blind Treatment Phase.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 66
Percent change | 4.10 (0.407) | 0.89 (0.413)
Statistical Analysis 1: Comparison: Denosumab 60 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [2.06 to 4.36]

2. Secondary Outcome: Mean Percent Change From Baseline in Lumbar Spine BMD at Month 1
Description: Mean percent change from Baseline in lumbar spine bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covariance (ANCOVA) model adjusting for treatment and Baseline BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Baseline=(measure at Month 1 - measure at Baseline) divided by the measure at Baseline * 100.
Time Frame: Baseline and Month 1
Population: ITTE Population
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 68 | 66
Percent change | 1.35 (0.375) | 0.62 (0.380)

3. Secondary Outcome: Mean Percent Change From Baseline in Total Hip, Femoral Neck, and Trochanter BMD at Month 1 and Month 6
Description: Mean percent change from Baseline in total hip, femoral neck, and trochanter bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covarience (ANCOVA) model adjusting for treatment and Baseline BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Baseline=(measure at Month 1/6 - measure at Baseline) divided by the measure at Baseline * 100.
Time Frame: Baseline, Month 1 and Month 6
Population: ITTE Population
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 64
Percent change
  Total hip, Month 1, n=67, 63 | 0.74 (0.238) | 0.05 (0.245)
  Total hip, Month 6, n=69, 64 | 2.23 (0.245) | 0.57 (0.254)
  Femoral neck, Month 1, n=67, 63 | 1.30 (0.344) | -0.04 (0.354)
  Fermoral neck, Month 6, n=69, 64 | 2.23 (0.330) | 0.84 (0.343)
  Trochanter, Month 1, n=67, 63 | 0.82 (0.380) | 0.39 (0.392)
  Trochanter, Month n =69, 64 | 2.66 (0.418) | 0.67 (0.434)

4. Secondary Outcome: Median Percent Change From Baseline in s-CTX and s-P1NP Biomarkers at Months 1, 3 and 6
Description: Serum carboxy-terminal cross-linking telopeptide of type I collagen (s-CTx) I and Serum procollagen type I N propeptide s (s-PINP) are used as serum biomarkers of bone resorption in the assessment of osteoporosis and is measured in units of micrograms (µg)/liters (L). Percentage change from Baseline=(measure at post-Baseline - measure at Baseline) divided by measure at Baseline * 100.
Time Frame: Baseline, Months 1, 3 and 6
Population: ITTE Population. Only participants at the specified time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 66
Percent change
  s-CTx, Month 1, n=69, 66 | -80.72 [-88.62 to -73.50] | -14.48 [-33.58 to -1.08]
  s-CTx, Month 3, n=68, 65 | -82.23 [-89.00 to -73.67] | -27.49 [-44.85 to -5.13]
  s-CTx, Month 6, n=60, 63 | -74.32 [-84.09 to -65.33] | -21.21 [-37.41 to 3.44]
  s-PINP, Month 1, n=69, 66 | -18.75 [-35.71 to -6.00] | -4.65 [-17.86 to 9.68]
  s-PINP, Month 3, n=68, 65 | -77.1 [-83.54 to -68.57] | -21.57 [-38.89 to -6.35]
  s-PINP, Month 6, n=60, 63 | -76.18 [-81.27 to -61.89] | -21.05 [-42.42 to -6.67]

5. Secondary Outcome: Number of Participants With Any Adverse Events (AE) or Any Serious Adverse Events (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury. Refer to the general Adverse AE/SAE module for a complete list of AEs and SAEs.
Time Frame: From Baseline up to Month 6
Population: Intent-to-Treat (ITT) Population: all participants who received one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 66
Participants
  Any AE | 38 | 32
  Any SAE | 7 | 2

6. Secondary Outcome: Change From Baseline in Albumin/Globulin Ratio and Blood Urea Nitrogen (BUN)/Creatinine Ratio at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Ratio
  Albumin/globulin ratio, n=60, 63 | 0.020 (0.1424) | 0.052 (0.1390)
  BUN/creatinine ratio, n=60, 63 | -7.917 (25.2917) | -4.063 (27.3436)

7. Secondary Outcome: Change From Baseline in Albumin, Hemoglobin, Mean Corpuscle Hemoglobin and Total Protein at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams (G)/Liter (L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Grams (G)/Liter (L)
  Albumin, n=60,63 | 0.217 (1.8964) | 0.365 (2.2598)
  Hemoglobin, n=59, 63 | 1.153 (5.8274) | 1.778 (5.6894)
  Mean corpuscle hemoglobin concentration, n=59, 63 | -5.186 (9.9264) | -6.857 (9.4593)
  Total protein, n=60, 63 | -0.050 (2.9939) | -0.127 (3.3864)

8. Secondary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Creatinine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed. .
Measure: Mean (Standard Deviation); unit: Internationational Units(IU)/Liter (L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Internationational Units(IU)/Liter (L)
  Alkaline phosphatase, n=60, 63 | -24.283 (15.9513) | -8.222 (11.2127)
  Alanine amino transferase, n=60, 63 | 2.117 (6.4047) | -0.397 (8.8035)
  Aspartate amino transferase, n=59, 63 | 1.034 (4.4527) | -0.032 (7.4962)
  Creatine kinase, n=60, 63 | 7.617 (51.6658) | 3.905 (31.2052)
  Gamma glutamyl transferase, n=60, 63 | -0.133 (8.4381) | -2.143 (7.9532)
  Lactate dehydraogenase, n=59, 63 | 6.119 (18.1156) | 3.889 (20.4979)

9. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Segmented Neutrophils, Platelet Count and White Blood Cell Count at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 58 | 63
10^9 cells per liter (GI/L)
  Basophils, n=58, 63 | -0.003 (0.0131) | -0.006 (0.0165)
  Eosinophils, n=58, 63 | -0.019 (0.1254) | -0.033 (0.1309)
  Lymphocytes, n=58, 63 | -0.047 (0.4096) | -0.206 (0.5930)
  Monocytes, n=58, 63 | -0.033 (0.1094) | -0.059 (0.1324)
  Segmented neutrophils, n=58, 63 | 0.114 (1.3382) | -0.213 (1.0934)
  Total neutrophils, n=58, 63 | 0.114 (1.3382) | -0.213 (1.0934)
  Platelet count, n=58, 63 | 1.621 (31.7881) | -6.190 (35.7874)
  White blood cell count, n=58, 63 | 0.014 (1.4026) | -0.517 (1.2003)

10. Secondary Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Creatinine and Uric Acid at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole/liter (UMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Micromole/liter (UMOL/L)
  Direct bilirubin, n=60, 63 | 0.300 (1.0301) | 0.222 (1.1974)
  Indirect bilirubin, n=60, 63 | 1.567 (3.4757) | 0.508 (3.5372)
  Total bilirubin, n=60, 63 | 1.867 (3.8947) | 0.730 (3.8404)
  Creatinine, n=60, 63 | 2.037 (6.4916) | 0.940 (5.1644)
  Uric acid, n=60, 63 | 11.500 (38.9622) | 0.159 (40.9757)

11. Secondary Outcome: Change From Baseline in Calcium Corrected, Calcium, Chloride, Glucose, Potassium, Magnesium, Sodium, Phosphorus Inorganic, Triglycerides, Urea/BUN, Very Low Density Lipoproteins (VLDL) Cholesterol Calculation at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole/Liter (MMOL/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Millimole/Liter (MMOL/L)
  Calcium (corrected), n=1, 1 | 0.110 (NA) — Only one participant was analyzed; therefore, the standard deviation was undefined. | 0.000 (NA) — Only one participant was analyzed; therefore, the standard deviation was undefined.
  Calcium, n=59, 63 | -0.020 (0.0890) | 0.002 (0.0768)
  Chloride, n=60, 63 | -0.200 (2.2981) | 0.444 (2.3264)
  Glucose, n=60, 63 | -0.873 (2.5458) | -0.567 (1.2118)
  Potassium, n=59, 63 | 0.000 (0.3900) | 0.060 (0.3476)
  Magnesium, n=60, 63 | 0.004 (0.0585) | 0.009 (0.0462)
  Sodium, n=60, 63 | -0.400 (2.1249) | 0.095 (1.9486)
  Phosphorus inorganic, n=60, 63 | -0.072 (0.1505) | -0.063 (0.1695)
  Triglycerides, n=60, 63 | -0.166 (0.7155) | -0.156 (0.6119)
  Urea/BUN, n=60, 63 | -0.258 (1.1878) | -0.119 (1.4134)
  VLDL cholesterol calculation, n=59, 63 | -0.098 (0.2844) | -0.072 (0.2810)

12. Secondary Outcome: Change From Baseline in Hematocrit at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of RBCs in blood
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 63
Proportion of RBCs in blood | 0.009 (0.0196) | 0.013 (0.0196)

13. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (PG)/cell
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 63
Picograms (PG)/cell | 0.068 (0.7111) | 0.146 (0.6696)

14. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (FL)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 63
Femtoliters (FL) | 1.695 (2.5000) | 2.397 (2.6368)

15. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 63
10^12 cells per liter (TI/L) | 0.025 (0.1844) | 0.037 (0.1920)

16. Secondary Outcome: Change From Baseline in Red Cell Distribution Width at Month 6
Description: Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage (%) of mean RBC volume
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 59 | 63
percentage (%) of mean RBC volume | 0.475 (1.0256) | 0.556 (0.9242)

17. Secondary Outcome: Number of Participants With a Change From Baseline in Vital Signs of Potential Clinical Concern at Month 6
Description: Vital Sign Changes from Baseline of potential clinical concern for Diastolic Blood Pressure (<50 or >120 Bits Per Minutes [bpm]), Systolic Blood Pressure (>170 Millimeters of Mercury [mmHg] or <100 mmHg) and Heart rate (>110 mmHg or <50 mmHg) are summarized. Change from Baseline was calculated as the Month 6 value minus the Baseline value.
Time Frame: Baseline and Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 60 | 63
Participants
  Diastolic blood pressure, Low, n=60, 63 | 0 | 2
  Systolic blood pressure, High, n=60, 63 | 1 | 2
  Systolic blood pressure, Low, n=60, 63 | 1 | 1
  Heart rate, High, n=60, 63 | 0 | 0
  Heart rate, Low, n=60, 63 | 0 | 0

18. Secondary Outcome: Number of Participants With Positive and Negative Results for Anti-body Formation to Denosumab
Description: Number of participants with positive and negative results for both neutralizing antibodies to denosumab, and for binding antibodies to denosumab at Month 6 was summarized.
Time Frame: Month 6
Population: ITT Population. Only participants at the specified time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg | Placebo
Number analyzed (Participants) | 69 | 66
Participants
  Neutralizing antibodies, Positive, n=0, 0 | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed. | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed.
  Neutralizing antibodies, Negative, n=0, 0 | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed. | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed.
  Binding antibodies, Positive, n=60, 63 | 0 | 0
  Binding antibodies, Negative, n=60, 63 | 60 | 63

19. Other Pre Specified Outcome: Mean Percent Change From Baseline in Lumbar Spine BMD at Month 12 for Participants Previously Randomized to Denosumab
Description: Mean percent change from Baseline in lumbar spine bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covariance (ANCOVA) model adjusting for treatment and Baseline BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Baseline=(measure at Month 12 - measure at Baseline) divided by the measure at Baseline * 100.
Time Frame: Baseline and Month 12
Population: Intent-to-Treat Open-Label (ITT-OL) Population: all participants from the ITT population in the Double-Blind Phase who continued into the Open-Label Extension Phase of the study and received denosumab at Month 6. Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg
Number analyzed (Participants) | 59
Percent change | 5.62 (3.776)

20. Other Pre Specified Outcome: Mean Percent Change From Month 6 in Lumbar Spine BMD at Month 12 for Participants Previously Randomized to Placebo
Description: Mean percent change from Month 6 in lumbar spine bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covariance (ANCOVA) model adjusting for treatment and Month 6 BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Month 6=(measure at Month 12 - measure at Month 6) divided by the measure at Month 6 * 100.
Time Frame: Month 6 and Month 12
Population: ITT-OL Population. Ony those participants with a value at Month 6 and Month 12 were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 59
Percent change | 2.67 (3.440)

21. Other Pre Specified Outcome: Mean Percent Change From Baseline in Total Hip, Femoral Neck, and Trochanter BMD at Month 12 for Participants Previously Randomized to Denosumab
Description: Mean percent change from Baseline in total hip, femoral neck, and trochanter bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covariance (ANCOVA) model adjusting for treatment and Baseline BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Baseline=(measure at Month 12 - measure at Baseline) divided by the measure at Baseline * 100.
Time Frame: Baseline and Month 12
Population: ITT-OL Population. Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg
Number analyzed (Participants) | 60
Percent change
  Total hip | 3.07 (2.476)
  Femoral neck | 3.39 (3.158)
  Trochanter | 3.39 (4.653)

22. Other Pre Specified Outcome: Mean Percent Change From Month 6 in Total Hip, Femoral Neck, and Trochanter BMD at Month 12 for Participants Previously Randomized to Placebo
Description: Mean percent change from Month 6 in total hip, femoral neck, and trochanter bone mineral density (BMD) was measured by the dual-energy x-ray absorptiometry (DXA) scanner. Analyses were performed using Analysis of Covariance (ANCOVA) model adjusting for treatment and Month 6 BMD for the skeletal site under consideration as a continuous covariate. Percentage change from Month 6=(measure at Month 12 - measure at Month 6) divided by the measure at Month 6 * 100.
Time Frame: Month 6 and Month 12
Population: ITT-OL Population. Ony those participants with a value at Month 6 and Month 12 were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 56
Percent change
  Total hip | 1.46 (1.701)
  Femoral neck | 1.12 (2.668)
  Trochanter | 2.13 (2.762)

23. Other Pre Specified Outcome: Median Percent Change From Baseline in s-CTX and s-P1NP Biomarkers at Month 12 for Participants Previously Randomized to Denosumab
Description: as for outcome 4
Time Frame: Baseline and Month 12
Population: ITT-OL Population. Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg
Number analyzed (Participants) | 57
Percent change
  s-CTx | -63.36 [-77.14 to -48.62]
  s-PINP | -78.00 [-84.31 to -66.67]

24. Other Pre Specified Outcome: Median Percent Change From Month 6 in s-CTX and s-P1NP Biomarkers at Month 12 for Participants Previously Randomized to Placebo
Description: Serum carboxy-terminal cross-linking telopeptide of type I collagen (s-CTx) I and Serum procollagen type I N propeptide s (s-PINP) are used as serum biomarkers of bone resorption in the assessment of osteoporosis and is measured in units of micrograms (µg)/liters (L). Percentage change from Month 6=(measure at Month 12 - measure at Month 6) divided by measure at Month 6 * 100.
Time Frame: Month 6 and Month 12
Population: ITT-OL Population. Ony those participants with a value at Month 6 and Month 12 were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60
Percent change
  s-CTx | -50.90 [-71.95 to -24.05]
  s-PINP | -66.67 [-76.82 to -55.65]

25. Other Pre Specified Outcome: Number of Participants With Any Adverse Events (AE) or Any Serious Adverse Events (SAE) During the Open-Label Extension Phase
Description: as for outcome 5
Time Frame: From Month 6 to Month 12
Population: ITT-OL Population
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Participants
  Any AE | 22 | 29
  Any SAE | 1 | 3

26. Other Pre Specified Outcome: Change From Baseline in Albumin/Globulin Ratio and Blood Urea Nitrogen (BUN)/Creatinine Ratio at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ITT-OL population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Ratio
  Albumin/globulin ratio, n=58, 60 | 0.016 (0.1473) | 0.032 (0.1621)
  BUN/creatinine ratio, n=58, 60 | -5.776 (24.4297) | 2.500 (27.7962)

27. Other Pre Specified Outcome: Change From Baseline in Albumin, Hemoglobin, Mean Corpuscle Hemoglobin and Total Protein at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams (G)/Liter (L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Grams (G)/Liter (L)
  Albumin, n=58, 60 | 0.293 (2.1110) | 0.450 (1.9866)
  Hemoglobin, n=56, 60 | 1.411 (5.7833) | 2.033 (6.0084)
  Mean corpuscle hemoglobin concentration, n=56, 60 | -5.679 (6.6143) | -6.650 (7.7587)
  Total protein, n=58, 60 | 0.224 (3.4946) | 0.267 (2.8216)

28. Other Pre Specified Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Creatinine Kinase, Gamma Glutamyl Transferase and Lactate Dehydrogenase at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Internationational Units(IU)/Liter (L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Internationational Units(IU)/Liter (L)
  Alkaline phosphatase, n=58, 60 | -25.603 (14.4780) | -23.767 (15.7570)
  Alanine amino transferase, n=58, 60 | 1.810 (7.9922) | -0.150 (8.9288)
  Aspartate amino transferase, n=58, 60 | 0.879 (6.4293) | -0.467 (6.2666)
  Creatine kinase, n=58, 60 | -4.534 (44.0690) | 4.500 (52.0731)
  Gamma glutamyl transferase, n=58, 60 | 0.4823 (6.9541) | -0.600 (9.4961)
  Lactate dehydraogenase, n=58, 60 | -0.552 (19.2237) | -1.217 (24.7243)

29. Other Pre Specified Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Segmented Neutrophils, Platelet Count and White Blood Cell Count at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
10^9 cells per liter (GI/L)
  Basophils, n=54, 59 | -0.004 (0.0164) | -0.002 (0.0148)
  Eosinophils, n=54, 59 | 0.024 (0.1489) | 0.019 (0.1860)
  Lymphocytes, n=54, 59 | 0.098 (0.4436) | -0.089 (0.5599)
  Monocytes, n=54, 59 | -0.009 (0.1053) | -0.039 (0.1443)
  Segmented neutrophils, n=54, 59 | 0.014 (1.1748) | -0.259 (1.2035)
  Total neutrophils, n=54, 59 | 0.014 (1.1748) | -0.259 (1.2035)
  Platelet count, n=55, 60 | -4.018 (34.8215) | -4.233 (37.7913)
  White blood cell count, n=54, 59 | 0.122 (1.1618) | -0.369 (1.3903)

30. Other Pre Specified Outcome: Change From Baseline in Direct Bilirubin, Indirect Bilirubin, Total Bilirubin, Creatinine and Uric Acid at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Micromole/liter (UMOL/L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Micromole/liter (UMOL/L)
  Direct bilirubin, n=58, 60 | 0.241 (1.3548) | 0.100 (1.2980)
  Indirect bilirubin, n=58, 60 | 1.034 (4.0391) | 0.800 (3.3385)
  Total bilirubin, n=58, 60 | 1.276 (4.6596) | 0.900 (3.5401)
  Creatinine, n=58, 60 | 0.948 (5.1157) | -0.015 (4.6216)
  Uric acid, n=58, 60 | 4.483 (41.3870) | 2.000 (44.0647)

31. Other Pre Specified Outcome: Change From Baseline in Calcium Corrected, Calcium, Chloride, Glucose, Potassium, Magnesium, Sodium, Phosphorus Inorganic, Triglycerides, Urea/BUN, Very Low Density Lipoproteins (VLDL) Cholesterol Calculation at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimole/Liter (MMOL/L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Millimole/Liter (MMOL/L)
  Calcium (corrected), n=0, 0 | NA (NA) — Zero participants was analyzed; therefore, the mean and the standard deviation were undefined. | NA (NA) — Zero participants was analyzed; therefore, the mean and the standard deviation were undefined.
  Calcium, n=58, 60 | -0.031 (0.0944) | -0.004 (0.0904)
  Chloride, n=58, 60 | 0.328 (2.5573) | 0.300 (2.4446)
  Glucose, n=58, 60 | -0.760 (2.9331) | -0.500 (1.2985)
  Potassium, n=58, 60 | 0.047 (0.4398) | 0.045 (0.3078)
  Magnesium, n=58, 60 | 0.009 (0.0679) | 0.004 (0.0514)
  Sodium, n=58, 60 | -0.172 (2.1532) | 0.067 (2.2986)
  Phosphorus inorganic, n=58, 60 | -0.153 (0.1530) | -0.094 (0.1981)
  Triglycerides, n=58, 60 | -0.144 (0.7716) | -0.033 (0.8449)
  Urea/BUN, n=58, 60 | -0.233 (1.2183) | 0.158 (1.5771)
  VLDL cholesterol calculation, n=58, 59 | -0.066 (0.3539) | -0.044 (0.3234)

32. Other Pre Specified Outcome: Change From Baseline in Hematocrit at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of RBCs in blood
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 56 | 60
Proportion of RBCs in blood | 0.010 (0.0182) | 0.014 (0.0185)

33. Other Pre Specified Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (PG)/cell)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 56 | 60
Picograms (PG)/cell) | -0.304 (0.7632) | -0.310 (0.5058)

34. Other Pre Specified Outcome: Change From Baseline in Red Blood Cell Count at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (TI/L)
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 56 | 60
10^12 cells per liter (TI/L) | 0.086 (0.1634) | 0.103 (0.1904)

35. Other Pre Specified Outcome: Change From Baseline in Red Cell Distribution Width at Month 12
Description: Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Mean (Standard Deviation); unit: percentage (%) of mean RBC volume
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 56 | 60
percentage (%) of mean RBC volume | 0.007 (0.7897) | 0.203 (0.8718)

36. Other Pre Specified Outcome: Number of Participants With a Change From Baseline in Vital Signs of Potential Clinical Concern at Month 12
Description: Vital Sign Changes from Baseline of potential clinical concern for Diastolic Blood Pressure (<50 or >120 Bits Per Minutes [bpm]), Systolic Blood Pressure (>170 Millimeters of Mercury [mmHg] or <100 mmHg) and Heart rate (>110 mmHg or <50 mmHg) are summarized. Change from Baseline was calculated as the Month 12 value minus the Baseline value.
Time Frame: Baseline and Month 12
Population: ITT-OL Population: Ony those participants with a value at Baseline and Month 12 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 58 | 61
Participants
  Diastolic blood pressure, High | 0 | 1
  Diastolic blood pressure, Low | 2 | 0
  Systolic blood pressure, High | 0 | 2
  Systolic blood pressure, Low | 0 | 2
  Heart rate, High | 0 | 0
  Heart rate, Low | 0 | 0

37. Other Pre Specified Outcome: Number of Participants With Positive and Negative Results for Anti-body Formation to Denosumab at Month 12
Description: Number of participants with positive and negative results for both neutralizing antibodies to denosumab, and for binding antibodies to denosumab at Month 12 was summarized.
Time Frame: Month 12
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | Denosumab 60 mg to Open-Label Denosumab 60mg | Placebo to Open-Label Denosumab 60 mg
Number analyzed (Participants) | 60 | 63
Participants
  Neutralizing antibodies, Positive, n=0, 0 | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed. | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed.
  Neutralizing antibodies, Negative, n=0, 0 | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed. | NA — There were no binding antibody confirmed positive tests; therefore, neutralizing antibody testing was not performed.
  Binding antibodies, Positive, n=58, 61 | 0 | 0
  Binding antibodies, Negative, n=58, 61 | 58 | 61

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study medication to the end of the Open-Label Phase (up to Month 12).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received one dose of study medication during the Double-Blind Treatment Phase, and for members of ITT-OL Population in the Open-Label Phase.
Groups:
- Randomized Phase: Denosumab 60 mg: Participants received a denosumab 60 milligrams (mg) single subcutaneous (SC) injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 International Units [IU]).
- Randomized Phase: Placebo: Participants received a matching placebo single SC injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU).
- Open Label Denosumab 60 mg (Previously Randomized Denosumab): Participants received a denosumab 60 milligrams (mg) single subcutaneous (SC) injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 International Units [IU]). At the end of the Double-Blind Treatment Phase, following completion of all Month 6 assessments, eligible participants entered the Open-Label Extension Phase and received a single SC injection of denosumab 60 mg and were followed up for an additional 6 months.
- Open Label Denosumab 60 mg (Previously Randomized Placebo): Participants received a matching placebo single SC injection at the start of the Double-Blind Treatment Phase. All participants received daily oral supplementation of elemental calcium (at least 1000 mg) and vitamin D (at least 400 IU). At the end of the Double-Blind Treatment Phase, following completion of all Month 6 assessments, eligible participants entered the Open-Label Extension Phase and received a single SC injection of denosumab 60 mg and were followed up for an additional 6 months.
Arm/Group | Randomized Phase: Denosumab 60 mg | Randomized Phase: Placebo | Open Label Denosumab 60 mg (Previously Randomized Denosumab) | Open Label Denosumab 60 mg (Previously Randomized Placebo)
Serious Adverse Events (participants affected / at risk) | 7/69 | 2/66 | 1/60 | 3/63
Other Adverse Events (participants affected / at risk) | 13/69 | 11/66 | 12/60 | 7/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: Denosumab 60 mg (N=69) | Randomized Phase: Placebo (N=66) | Open Label Denosumab 60 mg (Previously Randomized Denosumab) (N=60) | Open Label Denosumab 60 mg (Previously Randomized Placebo) (N=63)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Phase: Denosumab 60 mg (N=69) | Randomized Phase: Placebo (N=66) | Open Label Denosumab 60 mg (Previously Randomized Denosumab) (N=60) | Open Label Denosumab 60 mg (Previously Randomized Placebo) (N=63)
Constipation (Gastrointestinal disorders) | 5 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 8 | 6 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.